CLINICAL TRIAL: NCT05382494
Title: Efficacy of Intranasal Steroid for Children With Sleep-Disordered Breathing Non-Responsive to Initial Treatment With Intranasal Saline: A Randomized Trial
Brief Title: Intranasal Steroid as Medical Therapy For Sleep-Disordered Breathing in Children
Acronym: MIST+
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Murdoch Childrens Research Institute (Other)
Collaborators: Monash Health (Other); Royal Children's Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: RCH HREC 81746
Record Dates: First submitted 2022-05-16; First posted 2022-05-19 (Actual); Last update posted 2025-09-30 (Actual); Status verified 2025-09

CONDITIONS: Sleep Disorder; Breathing-Related; Snoring; Obstructive Sleep Apnea of Child; Sleep Disorders in Children; Tonsillar Hypertrophy; Adenoidal Disorder
MeSH Terms: conditions — Sleep Wake Disorders; Snoring | interventions — Mometasone Furoate; Nasal Sprays; Sodium Chloride

STUDY DESIGN:
Intervention Model Description: Multicentre, double-blind, randomised control trial
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The saline is the same colour and consistency to the active drug (intranasal steroid) and will have the same sensation when sprayed into the nostril. Randomisation will be stratified by site, Royal Children's Hospital (RCH) and Monash Health (MH), with permuted random block randomisation. An independent statistician in the Clinical Epidemiology and Biostatistics Unit (CEBU) at Murdoch Children's Research Institute (MCRI) will arrange the randomisation schedules, which will be given to the Clinical Trials Pharmacy at RCH and MH. This schedule will remain blinded to all other study staff.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intranasal Steroids (Experimental)
  Interventions: Drug: Mometasone Furoate 50mcg Nasal Spray
- Intranasal Saline (Placebo Comparator)
  Interventions: Drug: Sodium Chloride 0.9 % Nasal Spray

INTERVENTIONS:
Drug: Mometasone Furoate 50mcg Nasal Spray — Intranasal steroid (Mometasone Furoate 50mcg) one spray each nostril daily for 6 weeks
  Other Names: Sensease Nasal Allergy Relief Nasal Spray
  Arms: Intranasal Steroids
Drug: Sodium Chloride 0.9 % Nasal Spray — Intranasal saline spray (Sodium Chloride 0.9%) one spray each nostril daily for 6 weeks
  Other Names: Intranasal Saline Spray
  Arms: Intranasal Saline

SUMMARY:
MIST+ is studying a nasal spray to see if it will reduce the need for surgery for snoring. Children aged 3-12 are invited to take part. Snoring affects up to 10% of children and can cause sleeping problems and concentration or behavioural issues in the daytime. Currently the most common treatment for snoring is surgery to remove the tonsils and/or adenoids, however many children wait a long time to see a specialist. This research is trying to find if nasal sprays can help children with snoring, and whether this can reduce the need for surgery.

DETAILED DESCRIPTION:
MIST+ is a multi centre, double-blind, placebo controlled trial. Children 3-12 years of age, who do not respond to a run-in phase of 6 weeks of normal saline intranasal spray to treat sleep disordered breathing, will be randomised 1:1 to a treatment phase of either intranasal corticosteroid (investigational product) or normal saline (placebo). Participants will receive treatment for 6 weeks and receive follow up at at 12 weeks, 6, and 12 months.

ELIGIBILITY:
Inclusion Criteria:

Each participant must meet all of the following criteria to be enrolled in this trial:

* Is between the ages of 3 and 12 years inclusive at the time of randomisation
* Has symptoms of Sleep Disordered Breathing (SDB) as determined by a Brouillette score ≥ -1 on telehealth/phone screening
* Has a legally acceptable representative capable of understanding the informed consent document and providing consent on the participant's behalf.

Exclusion Criteria:

Participants meeting any of the following criteria will be excluded from the study:

* Has a BMI over the 97th centile for age and gender
* Has a history of tonsillectomy and/or adenoidectomy
* Has a prior diagnosis of craniofacial, neuromuscular, syndromic or defined genetic disorders
* Has a history of haemorrhagic diathesis or recurrent (daily) or severe epistaxis
* Has a history of nasal surgery or trauma which has not fully healed
* Has active tonsillitis or nasal infection (must be resolved prior to randomisation)
* Is assessed to have stertor (snoring) while awake at rest
* Has a known hypersensitivity to the study drug or its formulation
* Has used oral, intravenous, or intranasal steroids in the past 6 weeks. (Inhaled steroids for asthma will be allowed concomitantly during the study)
* Daily use of antihistamine or decongestant nasal sprays
* Is known to require systemic steroids prior to the completion of the study treatment phase
* Has had treatment with any other investigational drug within 6 months prior to randomisation
* Is unable to provide consent without the aid of an interpreter.
* In the opinion of the Investigator may be unable to follow the protocol

Ages: 3 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 130 (Actual)
Dates: Start 2022-12-05 (Actual); Primary Completion 2025-07-17 (Actual); Study Completion 2025-07-17 (Actual)

PRIMARY OUTCOMES:
The proportion of participants with resolution of significant Sleep Disordered Breathing (SDB) symptoms as defined by the parent completed Brouillette questionnaire </=-1 at 6 weeks | 6 weeks
  The Brouillette questionnaire is a validated symptom questionnaire that investigates the presence of respiratory sleep disorders and the frequency of apnoea and pathological snoring. Each item is scored from 0 to 3 (0 = absence of symptoms, 1 = occasional symptoms, 2 = frequent symptoms, and 3 = constant symptoms), and the overall score is directly proportional to disease severity.
  The proportion of participants in each treatment arm with resolution of symptoms at 6 weeks will be calculated with 95% confidence intervals (CIs). The treatment arms will be compared using a Mantel Haenszel chi-squared test.

SECONDARY OUTCOMES:
The proportion of participants with resolution of significant Sleep Disordered Breathing (SDB) symptoms as defined by the parent completed Brouillette questionnaire < -1 at 12 weeks | 12 weeks
  The Brouillette questionnaire is a validated symptom questionnaire that investigates the presence of respiratory sleep disorders and the frequency of apnoea and pathological snoring. Each item is scored from 0 to 3 (0 = absence of symptoms, 1 = occasional symptoms, 2 = frequent symptoms, and 3 = constant symptoms), and the overall score is directly proportional to disease severity.
  The proportion of participants in each treatment arm with resolution of symptoms at 12 weeks will be calculated with 95% confidence intervals (CIs). The treatment arms will be compared using a Mantel Haenszel chi-squared test.
An improvement of score in parent completed Pediatric Sleep Questionnaire-sleep disordered breathing subscale (PSQ-SDB subscale) at week 6 when compared with baseline measured at the start of the intervention period (week 0) | 6 weeks
  The Pediatric Sleep Questionnaire - sleep disordered breathing subscale is a validated questionnaire which contains 22 symptom items that ask about snoring frequency, loud snoring, observed apneas, difficulty breathing during sleep, daytime sleepiness, inattentive or hyperactive behaviour, and other paediatric Obstructive Sleep Apnoea (OSA) features. Responses are "yes" = 1, "no" = 0, and "don't know"=missing.
  The mean scores and 95% confidence intervals (CIs) in the two treatment arms will be calculated and the treatment arms will be compared using a linear regression adjusted for centre.
An improvement of score in parent completed Obstructive Sleep Apnoea-18 (OSA-18) questionnaire at week 6 when compared with baseline measured at the start of intervention period (week 0). | 6 weeks
  The Obstructive Sleep Apnoea-18 (OSA-18) questionnaire is a validated questionnaire and consists of 18 questions concerning sleep disturbances, physical symptoms, emotional distress, daytime function, and caregiver concerns.
  The mean scores and 95% confidence intervals (CIs) in the two treatment arms will be calculated and the treatment arms will be compared using a linear regression adjusted for centre.
An improvement of score in parent completed Pediatric Quality of Life Inventory (PedsQL) at week 6 when compared with baseline measured at the start of the intervention period (week 0). | 6 weeks
  The Pediatric Quality of Life Inventory (PedsQL) is a validated, standardised, generic assessment instrument that provides a modular approach to measure health related quality of life in healthy children and adolescents and those with acute and chronic disorders. This questionnaire consists of 23 items evaluating physical, emotional, social and scholastic functioning, and it integrates both generic core scales and disease-specific modules.
  The mean scores and 95% confidence intervals (CIs) in the two treatment arms will be calculated and the treatment arms will be compared using a linear regression adjusted for centre.
An improvement of score in parent completed Strengths and Difficulties Questionnaire (SDQ) at week 6 when compared with baseline measured at the start of the intervention period (week 0). | 6 weeks
  The Strengths and Difficulties Questionnaire (SDQ) is a validated brief behavioural screening questionnaire about 3-16 year olds. The mean scores and 95% confidence intervals (CIs) in the two treatment arms will be calculated and the treatment arms will be compared using a linear regression adjusted for centre.
An improvement of score in parent completed Glasgow Children's Benefit Inventory (GCBI) at week 6 when compared with baseline measured at the start of the intervention period (week 0). | 6 weeks
  The Glasgow Children's Benefit Inventory (GCBI) consists of 24 questions on the consequences of a specified intervention on various aspects of the day-to-day child life, without reference to any specific symptoms, and it can be apply to children of any age. The mean scores and 95% confidence intervals (CIs) in the two treatment arms will be calculated and the treatment arms will be compared using a linear regression adjusted for centre.
Proportion of parent responders who think their child needs surgery to remove their tonsils or adenoids (T&A) at 6 weeks | 6 weeks
  This will be measured by asking parents the following question on a parent assessment questionnaire developed for the study. "Do you think your child needs surgery to remove their tonsils or adenoids (T&A)?"
Proportion of parent responders who think their child needs surgery to remove their tonsils or adenoids (T&A) at 12 weeks | 12 weeks
  This will be measured by asking parents the following question on a parent assessment questionnaire developed for the study. "Do you think your child needs surgery to remove their tonsils or adenoids (T&A)?"
Proportion of parent responders who think their child needs surgery to remove their tonsils or adenoids (T&A) at 6 months | 6 months
  This will be measured by asking parents the following question on a parent assessment questionnaire developed for the study. "Do you think your child needs surgery to remove their tonsils or adenoids (T&A)?"
Proportion of parent responders who would be happy to proceed with tonsils and adenoids surgery (T&A) if recommended to them at 6 weeks | 6 weeks
  This will be measured by asking parents the following question on a parent assessment questionnaire developed for the study. "If T&A surgery were recommended to you now, would you be happy to proceed?"
Proportion of parent responders who would be happy to proceed with tonsils and adenoids (T&A) surgery if recommended to them at 12 weeks | 12 weeks
  This will be measured by asking parents the following question on a parent assessment questionnaire developed for the study: "If T&A surgery were recommended to you now, would you be happy to proceed?"
Proportion of parent responders who would be happy to proceed with tonsils and adenoids (T&A) surgery if recommended to them at 6 months | 6 months
  This will be measured by asking parents the following question on a parent assessment questionnaire developed for the study: "If T&A surgery were recommended to you now, would you be happy to proceed?"
Proportion of parent responders who would be happy to proceed with tonsils and adenoids (T&A) surgery if recommended to them at 12 months | 12 months
  This will be measured by asking parents the following question on a parent assessment questionnaire developed for the study: "If T&A surgery were recommended to you now, would you be happy to proceed?"
Proportion of parents who think their child still needs a review by a hospital specialist at 6 weeks | 6 weeks
  This will be measured by asking parents the following question on a parent assessment questionnaire developed for the study: "Do you think your child's symptoms need review by a hospital specialist?"
Proportion of parents who think their child still needs a review by a hospital specialist at 12 weeks | 12 weeks
  This will be measured by asking parents the following question on a parent assessment questionnaire developed for the study: "Do you think your child's symptoms need review by a hospital specialist?"
Proportion of parents who think their child still needs a review by a hospital specialist at 6 months | 6 months
  This will be measured by asking parents the following question on a parent assessment questionnaire developed for the study: "Do you think your child's symptoms need review by a hospital specialist?"
Proportion of parents who think their child still needs a review by a hospital specialist at 12 months | 12 months
  This will be measured by asking parents the following question on a parent assessment questionnaire developed for the study: "Do you think your child's symptoms need review by a hospital specialist?"
Proportion of parents who would be happy to have their child taken off the hospital clinic waiting list at 6 weeks | 6 weeks
  This will be measured by asking parents the following question on a parent assessment questionnaire developed for the study: "Would you be happy to have your child taken off the hospital clinic waiting list?"
Proportion of parents who would be happy to have their child taken off the hospital clinic waiting list at 12 weeks | 12 weeks
  This will be measured by asking parents the following question on a parent assessment questionnaire developed for the study: "Would you be happy to have your child taken off the hospital clinic waiting list?"
Proportion of parents who would be happy to have their child taken off the hospital clinic waiting list at 6 months | 6 months
  This will be measured by asking parents the following question on a parent assessment questionnaire developed for the study: "Would you be happy to have your child taken off the hospital clinic waiting list?"
Proportion of parents who would be happy to have their child taken off the hospital clinic waiting list at 12 months | 12 months
  This will be measured by asking parents the following question on a parent assessment questionnaire developed for the study: "Would you be happy to have your child taken off the hospital clinic waiting list?"
Parent satisfaction with run-in phase and treatment phase therapy as an alternative to tonsillectomy and/or adenoidectomy at 6 weeks (Likert Scale) | 6 weeks
  A study specific questionnaire using a 5 point Likert Scale will be used to evaluate parent satisfaction of ease of administration of drug, effectiveness of treatment, side effects. A higher score will indicate higher satisfaction. The mean scores and 95% confidence intervals in the two arms will be calculated and the treatment arms will compared using a linear regression adjusted for center.
Parent satisfaction with run-in phase and treatment phase therapy as an alternative to tonsillectomy and/or adenoidectomy at 12 weeks (Likert Scale) | 12 weeks
  A study specific questionnaire using a 5 point Likert Scale will be used to evaluate parent satisfaction of ease of administration of drug, effectiveness of treatment, side effects. A higher score will indicate higher satisfaction. The mean scores and 95% confidence intervals in the two arms will be calculated and the treatment arms will compared using a linear regression adjusted for center.
Progression to Tonsillectomy and/or Adenoidectomy for Sleep Disordered Breathing (SDB) defined by Ear Nose Throat (ENT) surgery at 6 months | 6 months
  Parents will be contacted by email with a short survey to record whether their child is either on a waitlist for ENT surgery or has undergone ENT surgery.
  The proportion of participants in each treatment arm who have progressed to Tonsillectomy and/or Adenoidectomy for SDB will be calculated with 95% confidence intervals. The treatment arms will be compared using a Mantel Haenszel chi-squared test.
Progression to Tonsillectomy and/or Adenoidectomy for Sleep Disordered Breathing defined by ENT surgery at 12 months | 12 months
  Parents will be contacted by email with a short survey to record whether their child is either on a waitlist for ENT surgery or has undergone ENT surgery.
  The proportion of participants in each treatment arm who have progressed to Tonsillectomy and/or Adenoidectomy for SDB will be calculated with 95% confidence intervals. The treatment arms will be compared using a Mantel Haenszel chi-squared test.
Progression to Tonsillectomy and/or Adenoidectomy for Sleep Disordered Breathing (SDB) based on symptoms of SDB reported in parent-completed Brouillette questionnaire at 6 months | 6 months
  The Brouillette questionnaire is a validated symptom questionnaire that investigates the presence of respiratory sleep disorders and the frequency of apnoea and pathological snoring. Each item is scored from 0 to 3 (0 = absence of symptoms, 1 = occasional symptoms, 2 = frequent symptoms, and 3 = constant symptoms), and the overall score is directly proportional to disease severity.
  The proportion of participants in each treatment arm with resolution of symptoms at 6 months will be calculated with 95% confidence intervals (CIs). The treatment arms will be compared using a Mantel Haenszel chi-squared test.
Progression to Tonsillectomy and/or Adenoidectomy for Sleep Disordered Breathing (SDB) based on symptoms of SDB reported in parent-completed Brouillette questionnaire at 12 months. | 12 months
  The Brouillette questionnaire is a validated symptom questionnaire that investigates the presence of respiratory sleep disorders and the frequency of apnoea and pathological snoring. Each item is scored from 0 to 3 (0 = absence of symptoms, 1 = occasional symptoms, 2 = frequent symptoms, and 3 = constant symptoms), and the overall score is directly proportional to disease severity.
  The proportion of participants in each treatment arm with resolution of symptoms at 12 months will be calculated with 95% confidence intervals (CIs). The treatment arms will be compared using a Mantel Haenszel chi-squared test.
Progression to Tonsillectomy and/or Adenoidectomy for Sleep Disordered Breathing (SDB) based on symptoms of SDB reported in parent-completed Pediatric Quality of Life Inventory (PedsQL) at 6 months | 6 months
  The Pediatric Quality of Life Inventory (PedsQL) is a validated, standardised, generic assessment instrument that provides a modular approach to measure health related quality of life in healthy children and adolescents and those with acute and chronic disorders. This questionnaire consists of 23 items evaluating physical, emotional, social and scholastic functioning, and it integrates both generic core scales and disease-specific modules.
  The proportion of participants in each treatment arm with resolution of symptoms at 6 months will be calculated with 95% confidence intervals (CIs). The treatment arms will be compared using a Mantel Haenszel chi-squared test.
Progression to Tonsillectomy and/or Adenoidectomy for Sleep Disordered Breathing (SDB) based on symptoms of SDB reported in parent-completed Pediatric Quality of Life Inventory (PedsQL) at 12 months | 12 months
  The Pediatric Quality of Life Inventory (PedsQL) is a validated, standardised, generic assessment instrument that provides a modular approach to measure health related quality of life in healthy children and adolescents and those with acute and chronic disorders. This questionnaire consists of 23 items evaluating physical, emotional, social and scholastic functioning, and it integrates both generic core scales and disease-specific modules.
  The proportion of participants in each treatment arm with resolution of symptoms at 12 months will be calculated with 95% confidence intervals (CIs). The treatment arms will be compared using a Mantel Haenszel chi-squared test.
Progression to Tonsillectomy and/or Adenoidectomy for Sleep Disordered Breathing (SDB) based on treatment for Sleep Disordered Breathing (SDB) at 6 months | 6 months
  Parents will be emailed a survey with the following questions about any treatment their child may have had for SDB
  1. Specialty of Dr seen and number of appointments
  2. Medical Treatment used, and duration of treatment The study team will describe additional treatment received by the treatment arm and investigate and describe any imbalance by the treatment arm.
Progression to Tonsillectomy and/or Adenoidectomy for Sleep Disordered Breathing (SDB) based on treatment for Sleep Disordered Breathing (SDB) at 12 months. | 12 months
  Parents will be asked the following questions about any treatment their child may have had for SDB
  1. Specialty of Dr seen and number of appointments
  2. Medical Treatment used, and duration he study team will describe additional treatment received by the treatment arm and investigate and describe any imbalance by the treatment arm. of treatment
Number of adverse events (AEs) throughout the treatment phase | 6 weeks
  Participants will also be asked questions about hospitalisation, accidents, new or changed medications. In addition AE's will be documented from physical examination findings, clinically significant lab results or other documents (including diaries where solicited AE's are prompted and correspondence from their primary care physician) that are relevant to participant safety. Adverse events and adverse reactions (non-serious or serious will be captured) The number of AEs will be summarised and listed in each of the treatment arms.
Number of adverse events (AEs) within the first week of the treatment | 1 week
  Participants will also be asked questions about hospitalisation, accidents, new or changed medications. In addition AE's will be documented from physical examination findings, clinically significant lab results or other documents (including diaries where solicited AE's are prompted and correspondence from their primary care physician) that are relevant to participant safety. Adverse events and adverse reactions (non-serious or serious will be captured) The number of AEs will be summarised and listed in each of the treatment arms.
Compliance of medical therapy measured by weight of sent and returned bottles of medication | -6 weeks and 6 weeks (start of run-in phase to end of treatment phase)
  Bottles will be weighed before they are given to participants and weighed when they are returned. The amount used will be calculated and used to determine if the participant was compliant with dosing. The amount of one spray of medication will be measured to allow for compliance to be calculated.
  Compliance with treatment will be calculated as the proportion of prescribed doses over 6 weeks that was consumed based on the weight of the bottles. The mean compliance will be summarised for the run-in period and both treatment arms. The proportion of participants with 80% and more compliance will be given for each treatment arm. The amount of one spray of medication will be measured to allow for compliance to be calculated.
Clinical factors at baseline that are associated with response to interventions, based on statistical analysis | 6 weeks
  Logistical regression models will be fitted to determine whether clinical factors at baseline or severity of SDB symptoms at baseline were associated with response to the intervention. Treatment arm, the symptom or factor of interest, and the interaction between the treatment arm and the symptom or factor will be included in this model. Symptoms or factors of interest include demographic factors, severity of SDB at baseline, history of atopy and history of tonsillitis.

CONTACTS AND LOCATIONS:
Overall Officials: Kirsten Perrett, Principal Investigator — Murdoch Children's Research Institute
Locations (2):
- Australia (2):
  - Monash Children's Hospital, Clayton, Victoria
  - Royal Children's Hospital / Murdoch Children's Research Institute, Parkville, Victoria

IPD SHARING:
Plan to Share IPD: Yes
The de-identified data set that will be collected for this analysis of the MIST+ trial will be available six months after publication of the primary outcome. The study protocol may be obtained from the Murdoch Children's Research Institute. Prior to releasing any data, the following are required: a data access agreement must be signed between relevant parties; the MIST+ trial investigators must see and approve the analysis plan describing how the data will be analysed; there must be an agreement around appropriate acknowledgment; and any additional costs involved must be covered.
  Should the study investigators be unavailable, this role is delegated to the Murdoch Children's Research Institute. Data will only be shared with a recognised research institute, which has approved the proposed analysis plan.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Six months after the publication of the primary outcome
Access Criteria: Prior to releasing any data, the following are required: a data access agreement must be signed between relevant parties; the MIST+ trial investigators must see and approve the analysis plan describing how the data will be analysed; there must be an agreement around appropriate acknowledgment; and any additional costs involved must be covered.
URL: https://www.mcri.edu.au/research/core-facilities-services/melbourne-children-trials-centre

REFERENCES:
- [Derived] Nixon GM, Anderson D, Baker A, Davidson A, Griffiths A, Grobler AC, Pinczower G, Rimmer J, Rose E, Selman CJ, Simpson CM, Vandeleur M, Perrett KP. Intranasal Treatments for Children With Sleep-Disordered Breathing: The MIST+ Randomized Clinical Trial. JAMA Pediatr. 2026 Jan 20:e255717. doi: 10.1001/jamapediatrics.2025.5717. Online ahead of print. PMID 41557344